CLINICAL TRIAL: NCT04213079
Title: Treatments of Mal de Debarquement Syndrome (MdDS) by Habituation of Velocity Storage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Sergei Yakushin, Associate Professor, Neurology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO-19-0348; 1R21DC018390-01 (NIH)
Record Dates: First submitted 2019-12-23; First posted 2019-12-30 (Actual); Results first posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Mal de Debarquement Syndrome (MdDS)
Keywords: Mal de Debarquement Syndrome; Motion Sickness; body rocking; body swaying; Habituation of velocity storage
MeSH Terms: conditions — Mal de debarquement; Motion Sickness; Stereotypic Movement Disorder

STUDY DESIGN:
Intervention Model Description: In this project, 50 motion triggered MdDS patients with otherwise normal vestibular and neurological functions will be randomly assigned into two groups, one to be treated by velocity storage habituation and the other by readaptation. Patients will be followed up for 6 months. Based on the preliminary data, we expect both groups to yield similar initial success rates for symptom improvement.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Vestibulo-ocular reflex (VOR) (Experimental): Treatment by re-adaptation of the vestibulo-ocular reflex (VOR) for participants with motion triggered MdDS
  Interventions: Device: re-adaptation of the vestibulo-ocular reflex
- Habituation of velocity storage (Experimental): Participants with motion triggered MdDS
  Interventions: Device: Habituation of velocity storage of the vestibulo-ocular reflex

INTERVENTIONS:
Device: re-adaptation of the vestibulo-ocular reflex — The VOR will be readapted by activating velocity storage with full-field optokinetic motion at 5°/s in a set direction while the head is oscillated with a set frequency and direction. The readaptation training will be conducted in repeated modules, each lasting for 1-5 min. The expected duration of daily sessions varies from 30 to 90 min. A day's session will be terminated if patient no longer feel symptoms of MdDS.
  Arms: Vestibulo-ocular reflex (VOR)
Device: Habituation of velocity storage of the vestibulo-ocular reflex — The central (velocity storage) time constant will be reduced by inducing cancellation of two velocity storage-mediated responses: OKN and the VOR. Sinusoidal rotation at 0.017 Hz (1 revolution/min) in darkness advances the slow phase eye velocity of the VOR by 32º. In contrast, the OKN at this frequency has no phase advancement. Thus, to counteract the VOR by OKN, the optokinetic stimulus should be set to 32º phase advance the out of phased head rotation stimulus. Since the conflict stimulus is expected to be overwhelming to patients at higher chair velocities, subjects will be first trained with a 10°/s stimulus. In a previous study, no complaints were reported when subjects were tested at such low velocities. Preliminary testing show signs of symptom improvement when the peak velocity reached 30°/s to 40°/s.
  Arms: Habituation of velocity storage

SUMMARY:
Mal de Debarquement Syndrome (MdDS) is an under-recognized but nevertheless common balance disorder, which in most cases occurs after exposure to prolonged passive motion. The current treatment approaches focus on reducing symptoms, but they can be retriggered. This project aims to shift the focus of MdDS treatment to permanently eliminating the symptom trigger while also minimizing symptoms.

DETAILED DESCRIPTION:
Mal de Debarquement Syndrome (MdDS) is an under-recognized but nevertheless common balance disorder, primarily manifested by constant self-motion sensations consisting of rocking/swaying or gravitational pull of the body, which are accompanied by fatigue, migraine, hypersensitivity to light/noise/crowds, visually induced dizziness, and cognitive dysfunctions. As the name implies ("disembarkation sickness"), in most cases MdDS occurs after exposure to prolonged passive motion, specified as motion-triggered (MT) MdDS. However, the symptoms of MdDS can also occur without a motion trigger, termed as spontaneous MdDS. MdDS is debilitating and entails various mental health issues, such as suicidal thoughts, depression, and anxiety. Treatments for this disorder are still limited, as the specific underlying pathophysiology remains unclear. Recently, the team developed the first treatment method that can safely and effectively ease MdDS symptoms in the majority of patients via readaptation of the vestibulo-ocular reflex (VOR). The hypothesis underlying this treatment is that MdDS is caused by maladaptation of the functional component of the VOR called velocity storage, whose readaptation can be stimulated by exposure to whole-field visual motion coupled with head tilts. Over the past several years, more than 500 patients from around the world have been treated with this method. The success rate immediately after this treatment is 75% for MT MdDS, but some patients report return of symptoms after subsequent flights or prolonged car rides. Thus, the effectiveness of the current MdDS treatment protocol can depend on a serious practical limitation of needing to permanently avoid transportation. Building on the previous hypothesis of velocity storage maladaptation, the study team currently hypothesizes that another method, based on the reduction (habituation) of the velocity storage, can also resolve MdDS symptoms. Velocity storage can be greatly habituated within 4-5 days using a protocol previously developed in the study team's laboratory to reduce susceptibility to motion sickness. Preliminary data support the application of this protocol to MdDS. Moreover, since animal-based research suggests that velocity storage habituation is permanently retained, the study team further hypothesizes that this new treatment method yields robust long-term outcomes. In this project, 50 MT MdDS patients with otherwise normal vestibular and neurological functions will be randomly assigned into two groups, one to be treated by velocity storage habituation and the other by readaptation. Patients will be followed up for 6 months. Based on the preliminary data, the study team expects both groups to yield similar initial success rates for symptom improvement. However, the study team expects the group undergoing the habituation protocol to better retain the initial treatment impact in the long term. This project will significantly impact the MdDS treatment practice. The current approach focuses on reducing symptoms, but they can be retriggered by another prolonged exposure to passive motion. The habituation approach on the other hand focuses on permanently minimizing the symptom trigger while also minimizing symptoms. This project will also increase the current understanding of recurrent MdDS.

ELIGIBILITY:
Inclusion Criteria:

- Age 18-78.

Exclusion Criteria:

- Patient with serious spinal, neck and legs injuries will be excluded, since postural ability is essential for both treatments.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergei Yakushin, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Vestibular Testing Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal to achieve aims in the approved proposal.

REFERENCES:
- [Background] Dai M, Cohen B, Cho C, Shin S, Yakushin SB. Treatment of the Mal de Debarquement Syndrome: A 1-Year Follow-up. Front Neurol. 2017 May 5;8:175. doi: 10.3389/fneur.2017.00175. eCollection 2017. PMID 28529496
- [Background] Yakushin SB, Palla A, Haslwanter T, Bockisch CJ, Straumann D. Dependence of adaptation of the human vertical angular vestibulo-ocular reflex on gravity. Exp Brain Res. 2003 Sep;152(1):137-42. doi: 10.1007/s00221-003-1543-0. Epub 2003 Jul 17. PMID 12879171
- [Background] Eron JN, Cohen B, Raphan T, Yakushin SB. Adaptation of orientation of central otolith-only neurons. Ann N Y Acad Sci. 2009 May;1164:367-71. doi: 10.1111/j.1749-6632.2009.03848.x. PMID 19645928
- [Background] Yakushin SB, Xiang Y, Cohen B, Raphan T. Dependence of the roll angular vestibuloocular reflex (aVOR) on gravity. J Neurophysiol. 2009 Nov;102(5):2616-26. doi: 10.1152/jn.00245.2009. Epub 2009 Aug 19. PMID 19692515
- [Background] Kolesnikova OV, Raphan T, Cohen B, Yakushin SB. Orientation adaptation of eye movement-related vestibular neurons due to prolonged head tilt. Ann N Y Acad Sci. 2011 Sep;1233:214-8. doi: 10.1111/j.1749-6632.2011.06176.x. PMID 21950996
- [Background] Mucci V, Canceri JM, Brown R, Dai M, Yakushin SB, Watson S, Van Ombergen A, Jacquemyn Y, Fahey P, Van de Heyning PH, Wuyts F, Browne CJ. Mal de Debarquement Syndrome: A Retrospective Online Questionnaire on the Influences of Gonadal Hormones in Relation to Onset and Symptom Fluctuation. Front Neurol. 2018 May 24;9:362. doi: 10.3389/fneur.2018.00362. eCollection 2018. PMID 29910765
- [Background] Mucci V, Canceri JM, Brown R, Dai M, Yakushin S, Watson S, Van Ombergen A, Topsakal V, Van de Heyning PH, Wuyts FL, Browne CJ. Mal de Debarquement Syndrome: a survey on subtypes, misdiagnoses, onset and associated psychological features. J Neurol. 2018 Mar;265(3):486-499. doi: 10.1007/s00415-017-8725-3. Epub 2018 Jan 5. PMID 29305644
- [Background] Dai M, Cohen B, Smouha E, Cho C. Readaptation of the vestibulo-ocular reflex relieves the mal de debarquement syndrome. Front Neurol. 2014 Jul 15;5:124. doi: 10.3389/fneur.2014.00124. eCollection 2014. PMID 25076935
- [Background] Cohen B, Dai M, Yakushin SB, Cho C. The neural basis of motion sickness. J Neurophysiol. 2019 Mar 1;121(3):973-982. doi: 10.1152/jn.00674.2018. Epub 2019 Jan 30. PMID 30699041
- [Background] Dai M, Raphan T, Cohen B. Prolonged reduction of motion sickness sensitivity by visual-vestibular interaction. Exp Brain Res. 2011 May;210(3-4):503-13. doi: 10.1007/s00221-011-2548-8. Epub 2011 Feb 2. PMID 21287155
- [Background] Cohen B, Dai M, Yakushin SB, Raphan T. Baclofen, motion sickness susceptibility and the neural basis for velocity storage. Prog Brain Res. 2008;171:543-53. doi: 10.1016/S0079-6123(08)00677-8. PMID 18718351
- [Background] Cohen B, Yakushin SB, Cho C. Hypothesis: The Vestibular and Cerebellar Basis of the Mal de Debarquement Syndrome. Front Neurol. 2018 Feb 5;9:28. doi: 10.3389/fneur.2018.00028. eCollection 2018. PMID 29459843
- [Background] Yakushin SB, Raphan T, Cohen B. Coding of Velocity Storage in the Vestibular Nuclei. Front Neurol. 2017 Aug 16;8:386. doi: 10.3389/fneur.2017.00386. eCollection 2017. PMID 28861030
- [Background] Eron JN, Ogorodnikov D, Horn AKE, Yakushin SB. Adaptation of spatio-temporal convergent properties in central vestibular neurons in monkeys. Physiol Rep. 2018 Sep;6(17):e13750. doi: 10.14814/phy2.13750. PMID 30178612
- [Background] Eron JN, Cohen B, Raphan T, Yakushin SB. Adaptation of orientation vectors of otolith-related central vestibular neurons to gravity. J Neurophysiol. 2008 Sep;100(3):1686-90. doi: 10.1152/jn.90289.2008. Epub 2008 May 21. PMID 18497367
- See also: Guidelines for patients coming for the treatment. Available treatment announcements — http://mdds.nyc/
- Available data/document: Study Protocol — http://mdds.nyc/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from April 2020 -July 2022 with first enrollment in June 2020; Patient volunteers with MdDS were recruited through various sources of referral and announcements posted on the Internet, including ClinicalTrials.gov (NCT04213079). Applicants seeking treatment were screened with an intake form, and each candidate's diagnosis of MdDS with an associable motion trigger was confirmed by a board-certified physician through a telephone interview when necessary.
Period: Overall Study
Arm/Group | Vestibulo-ocular Reflex (VOR) | Habituation of Velocity Storage
Started | 24 | 23
Completed | 24 | 21
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vestibulo-ocular Reflex (VOR) | Habituation of Velocity Storage | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (13.9) | 46.7 (14.2) | 47.1 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 16 | 38
  Male | 2 | 5 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subjective Symptoms Self-report of Overall Severity
Description: The overall severity of MdDS-related symptoms was subjectively reported on a single 11-point scale of 0-10, where the score 0 indicated no symptoms and 10 the most difficult of combined symptoms that the patient subject could imagine. Higher score indicates poorer health outcomes. Among the symptoms to consider were: brain fog, head pressure, fullness of ear, heavy head, headache, nausea, blurry vision, fatigue, sensitivity to fluorescent lights, scrolling of computer screen, sensitivity to smell, sensitivity to noise, walking on trampoline, sensation of gravitational pull up or down. Subjects were trained to estimate the level of symptoms to minimize inconsistency.
Time Frame: During treatment (Day 1), Day 5, and 6 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vestibulo-ocular Reflex (VOR) | Habituation of Velocity Storage
Number analyzed (Participants) | 24 | 21
score on a scale
  Day 1 | 5.2 (1.9) | 5.2 (1.9)
  Day 5 | 3.2 (2.1) | 2.1 (1.7)
  6 month follow up | 2.9 (2.0) | 3.4 (2.2)

2. Secondary Outcome: Visual Vertigo Analogue Scale (VVAS)
Description: Visual Vertigo Analogue Scale. There are 9 separate visual analogue scales to rate intensity of visual vertigo provoking situation. Each scale is on a 0-10 cm line. Full scale from 0-10. Higher score represents more dizziness.
Time Frame: Baseline and 6 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vestibulo-ocular Reflex (VOR) | Habituation of Velocity Storage
Number analyzed (Participants) | 24 | 21
score on a scale
  Baseline | 4.8 (2.0) | 4.4 (2.3)
  6 month follow up | 2.5 (2.1) | 2.6 (2.2)

3. Secondary Outcome: Dizziness Handicap Inventory (DHI) Questionnaire
Description: Physical, emotional, and functional disability related to MdDS will be assessed with DHI. DHI is a 25-item self report questionnaire, total score range from 0 to 100, with higher score indicating more perceived disability.
Time Frame: Baseline and 6 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vestibulo-ocular Reflex (VOR) | Habituation of Velocity Storage
Number analyzed (Participants) | 24 | 21
score on a scale
  Baseline | 52.1 (17.3) | 47.2 (16.1)
  6 month follow up | 35.3 (19.5) | 32.1 (18.6)

4. Secondary Outcome: VOR Direct Pathway Gain
Description: The vestibulo-ocular reflex (VOR) is a class of reflex eye movement that counters head movement to stabilize vision. A perfect stabilization occurs when the velocity of the retinal image slip is zero, i.e. when the ratio, or gain, of the eye rotation speed to the head rotation speed is one. The VOR is a fast reflex whose direct pathway consists of a three-neuron arc, but also has parallel, indirect pathways that allow integration of signals from the peripheral vestibular organs with those of other sensory modalities such as vision and proprioception to modulate the eye movement response. The gain of the direct VOR pathway is the ratio of the eye rotation speed to the head rotation speed at the onset of head rotation, and is a unitless measure.
Time Frame: Baseline and Day 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Vestibulo-ocular Reflex (VOR) | Habituation of Velocity Storage
Number analyzed (Participants) | 24 | 21
ratio
  Baseline | 0.53 (0.13) | 0.42 (0.10)
  6 month follow up | 0.45 (0.14) | 0.47 (0.08)

5. Secondary Outcome: VOR Indirect Pathway Time Constant
Description: The velocity storage mechanism is an indirect component of the VOR that facilitates the reflex by storing and releasing signals related to head rotation, for example by prolonging the eye movement response beyond the peripheral vestibular activity during head movement and generating similar eye movement response to rotational cues provided by other sensory modalities. The time constant of this indirect VOR pathway is the rate of charging/discharging in the exponential ideation of its behavior, measured in seconds, estimated from the profile of eye rotation speed during prolonged whole-body rotation that is the combination of the contributions from the direct and indirect pathways.
Time Frame: Baseline and Day 5
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Vestibulo-ocular Reflex (VOR) | Habituation of Velocity Storage
Number analyzed (Participants) | 24 | 21
seconds
  Baseline | 16.6 (3.9) | 15.0 (4.0)
  Day 5 | 16.0 (5.4) | 15.6 (4.5)

6. Secondary Outcome: VOR Indirect Pathway Coupling Gain
Description: The gain of the indirect VOR pathway is the term that determines the contribution of velocity storage to the profile of eye rotation speed during prolonged whole-body rotation. The measure is normalized to the head rotation velocity and is thus unitless.
Time Frame: Baseline and Day 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Vestibulo-ocular Reflex (VOR) | Habituation of Velocity Storage
Number analyzed (Participants) | 24 | 21
ratio
  Baseline | 0.102 (0.022) | 0.093 (0.030)
  Day 5 | 0.080 (0.033) | 0.099 (0.027)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Vestibulo-ocular Reflex (VOR) | Habituation of Velocity Storage
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 0/24 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT04213079/Prot_000.pdf
  • Informed Consent Form (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT04213079/ICF_001.pdf